CLINICAL TRIAL: NCT02257723
Title: The Effect of Integrated CAM Treatment in Patients Hospitalized at a Korean Medicine Hospital
Brief Title: The Effect of Integrated CAM Treatment in Hospitalized Patients
Status: Recruiting | Type: Observational
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2012-03
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain; Neck Pain; Knee Pain; Shoulder Pain; Intervertebral Disc Herniation; Spinal Stenosis
Keywords: Inpatient care; Complementary and alternative medicine; Integrated medicine
MeSH Terms: conditions — Low Back Pain; Neck Pain; Shoulder Pain; Intervertebral Disc Displacement; Spinal Stenosis | interventions — Phytotherapy; Acupuncture Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Herbal medicine — Herbal medicine was taken 3 times daily in dried powder (2g) and water-base decoction form (120ml) (Ostericum koreanum, Eucommia ulmoides, Acanthopanax sessiliflorus, Achyranthes bidentata, Psoralea corylifolia, Peucedanum japonicum, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, and Atractylodes japonica).
  Other Names: Traditional herbal medicine
Procedure: Acupuncture — Acupuncture treatment was administered 1-2 times daily using mainly Ah-shi points and local acupuncture points.
Procedure: Pharmacopuncture — Select ingredients similar to those included in the oral herbal medicine (Ostericum koreanum, Eucommia ulmoides, Acanthopanax Sessiliflorus, Achyranthes bidentata, Psoralea corylifolia, Peucedanum japonicum, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, and Atractylodes japonica) were freeze dried into powder form after decoction, then diluted in normal saline and adjusted for acidity and pH to be used in injections. The pharmacopuncture injections were injected once daily to the amount of 1 cc and Ah-shi points and local acupuncture points (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
Procedure: Bee venom pharmacopuncture — Bee venom pharmacopuncture was applied after confirming a negative reaction to the hypersensitivity skin test. Diluted bee venom (saline:bee venom ratio, 10,000:1) was injected at 4-5 acupoints at the physician's discretion. Each acupuncture point was injected with approximately 0.2 cc to a total of 0.5-1 cc using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
Procedure: Chuna manipulation — Chuna was administered 3-5 times a week. Chuna is a Korean version of spinal manipulation that incorporates conventional spinal manipulation techniques for mobilization involving high-velocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement.

SUMMARY:
This study investigates the effect of hospital-based intensive non-surgical treatment in musculoskeletal patients admitted to an integrated hospital that offers both complementary and alternative medicine (CAM) and conventional medicine treatment.

DETAILED DESCRIPTION:
This study investigates the effect of hospital-based intensive non-surgical treatment in musculoskeletal patients admitted to an integrated hospital that offers both complementary and alternative medicine (CAM) and conventional medicine treatment.

Inpatients received treatment according to a CAM treatment protocol (herbal medicine, acupuncture, bee venom pharmacopuncture, and Chuna manipulation) and conventional medicine treatment as needed. The main outcome measures were the duration of pain, NRS of back pain, radiating leg pain, neck pain, radiating arm pain, knee pain, shoulder pain, previous surgery, previous interventions (injections), Oswestry Disability Index (ODI), Vernon-Mior Neck Disability Index, the Korean Western Ontario McMaster Index, Shoulder Pain and Disability Index, range of motion (ROM), Straight leg raise test (SLR), alcohol use, smoking at admission, 2 weeks, and discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized due to spine or joint diseases

Exclusion Criteria:

* Main complaint other than back pain, radiating leg pain, neck pain, radiating arm pain, knee pain or shoulder pain
* Cause of pain non-related to spine, joint or soft tissue; for example, spinal tumors, pregnancy, urolithiasis, etc.
* Refusal to provide the information needed for clinical research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Musculoskeletal patients admitted to an integrated hospital that offers both complementary and alternative medicine (CAM) and conventional medicine treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
NRS of low back pain (LBP) | Admission (baseline), 2 weeks, Discharge
  The patients were asked to quantify their current LBP, setting no pain as 0 and the most severe pain that they could possibly imagine as 10.
NRS of radiating leg pain | Admission (baseline), 2 weeks, Discharge
  The patients were asked to quantify their current leg pain, setting no pain as 0 and the most severe pain that they could possibly imagine as 10.
NRS of neck pain | Admission (baseline), 2 weeks, Discharge
  The patients were asked to quantify their current neck pain, setting no pain as 0 and the most severe pain that they could possibly imagine as 10.
NRS of radiating arm pain | Admission (baseline), 2 weeks, Discharge
  The patients were asked to quantify their current radiating arm pain, setting no pain as 0 and the most severe pain that they could possibly imagine as 10.
NRS of knee pain | Admission (baseline), 2 weeks, Discharge
  The patients were asked to quantify their current knee pain, setting no pain as 0 and the most severe pain that they could possibly imagine as 10.
NRS of shoulder pain | Admission (baseline), 2 weeks, Discharge
  The patients were asked to quantify their current shoulder pain, setting no pain as 0 and the most severe pain that they could possibly imagine as 10.
Oswestry disability index (ODI) | Admission (baseline), 2 weeks, Discharge
  The ODI is a survey assessing the patients' degree of functional disability in daily life consisting of 10 questions with 6 choices each corresponding to 0-5 points. The scores for each item are added, divided by 50, then multiplied by 100 to calculate the degree of disability. The Korean version of the ODI of which the reliability and validity have been verified through the research of Jeon et al. was used in this study.
Vernon-Mior Neck Disability Index (NDI) | Admission (baseline), 2 weeks, Discharge
  NDI is a survey for evaluating disabilities that can be caused by neck pain in daily life performance. It consists of a total of 50 points by selecting a number from 0 to 5 for each item in 10 questions. The higher the score, the greater the daily disability.
The Korean Western Ontario McMaster Index | Admission (baseline), 2 weeks, Discharge
  WOMAC is one of the most widely used indicators of the overall joint function score of the knee joint. A tool for evaluating disorders related to osteoarthritis of the lower extremities, including joints or knee joints.
  WOMAC consists of a total of 24 questions and three subscales. It consists of 5 questions about pain, 2 questions about stiffness, and 17 questions about difficulty in performing daily life related to the rest of the physical functions, so it is designed to measure the overall functional state of the joint.
Shoulder Pain and Disability Index | Admission (baseline), 2 weeks, Discharge
  SPADI is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.

SECONDARY OUTCOMES:
Physical and neurological examinations | Admission (baseline), 2 weeks, Discharge
  The range of flexion and extension was assessed to objectively measure mobility, and straight leg raising (SLR), sensory function, muscle strength, and deep tendon reflex tests were conducted for neurological assessment.

OTHER OUTCOMES:
Other baseline variables | Admission (baseline)
  The duration of pain, previous surgery, previous interventions (injections), alcohol use, smoking

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, PhD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

REFERENCES:
- [Derived] Kim MH, Lee YJ, Shin JS, Lee J, Jeong H, Kim MR, Park SM, Go U, Kim SM, Kim JY, Hwang DG, Ha IH. The Long-Term Course of Outcomes for Lumbar Intervertebral Disc Herniation following Integrated Complementary and Alternative Medicine Inpatient Treatment: A Prospective Observational Study. Evid Based Complement Alternat Med. 2017;2017:5239719. doi: 10.1155/2017/5239719. Epub 2017 Aug 27. PMID 28928789
- [Derived] Baek SH, Oh JW, Shin JS, Lee J, Lee YJ, Kim MR, Ahn YJ, Choi A, Park KB, Shin BC, Lee MS, Ha IH. Long term follow-up of cervical intervertebral disc herniation inpatients treated with integrated complementary and alternative medicine: a prospective case series observational study. BMC Complement Altern Med. 2016 Feb 4;16:52. doi: 10.1186/s12906-016-1034-z. PMID 26850111